CLINICAL TRIAL: NCT02288169
Title: Patient Outcomes of a Self-care Management Approach to Cancer Symptoms: A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: USflorida
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
Keywords: Symptom management; palliative care
MeSH Terms: conditions — Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- COPE (Experimental): The experimental group will receive usual care plus the COPE intervention. This group will receive 3 individual intervention sessions. During the first intervention visit at the cancer center, the COPE group will be taught the COPE intervention in a session focusing on the patient's self-identified most bothersome symptom. Role modeling and additional instruction will be provided via video, and patients will receive the Home Care Guide for Cancer and a copy of the video to take home. Three subsequent visits with the patient during regularly scheduled clinic visits will reinforce the principles of COPE and the use of the Home Care Guide, and will help patients apply this approach to managing other symptoms. In addition they will get 2 phone calls encouraging them to apply COPE.
  Interventions: Behavioral: COPE
- Support (Sham Comparator): The attention control group will receive supportive visits from the research team at the cancer center and subsequent meetings during clinic visits plus 2 subsequent supportive telephone calls, matched for time with COPE participants.
  Interventions: Behavioral: Support/Attention Control
- Control (No Intervention): The control group will receive usual care and no additional attention from our interventionists.

INTERVENTIONS:
Behavioral: COPE — We propose to test a brief, effective intervention with outpatients in a cancer center, with the goal of teaching patients symptom management skills for self-identified symptoms of highest priority to patients. The proposed randomized clinical trial will test the efficacy of the COPE intervention with patients with symptoms of moderate to high intensity, distress, frequency or interference with their lives as a result of their cancer.
  Arms: COPE
Behavioral: Support/Attention Control — The attention control group will receive supportive visits from the research team at the cancer center and subsequent meetings during clinic visits plus 2 subsequent supportive telephone calls
  Arms: Support

SUMMARY:
Regardless of their treatment, cancer patients endure a variety of difficult symptoms during their disease with averages ranging from 7 to 14 symptoms each. Cancer-related symptoms, especially when symptoms are very intense, distressing, frequent, or interfere with daily activities, can lead to depression, anxiety, and diminished quality of life. Improving their ability to self-manage difficult symptoms has the potential to diminish suffering, improve quality of life and decrease emergency room visits and associated costs. The investigators propose to test a brief, effective intervention with outpatients in a cancer center, with the goal of teaching patients symptom management skills for self-identified symptoms of highest priority to patients. Objective: The proposed randomized clinical trial will test the efficacy of the COPE intervention with patients with symptoms of moderate to high intensity, distress, frequency or interference with their lives as a result of their cancer. Method: The investigators will seek 300 completed subjects, outpatients with breast, colorectal, lung, and prostate cancers. Patients will be randomized into three groups. Group III, the experimental group, will receive usual care plus the COPE intervention. This group will receive 3 individual intervention sessions. During the first intervention visit at the cancer center, the COPE group will be taught the COPE intervention in a session focusing on the patient's self-identified most bothersome symptom. Role modeling and additional instruction will be provided via video, and patients will receive the Home Care Guide for Cancer and a copy of the video to take home. Three subsequent visits with the patient during regularly scheduled clinic visits will reinforce the principles of COPE and the use of the Home Care Guide, and will help patients apply this approach to managing other symptoms. In addition they will get 2 phone calls encouraging them to apply COPE. Group II, the attention control group, will receive supportive visits from the research team at the cancer center and subsequent meetings during clinic visits plus 2 subsequent supportive telephone calls, matched for time with COPE participants. Group I, the control group receiving usual care, will receive no additional attention from our interventionists. Data will be collected weekly for 9 weeks about symptoms (intensity, frequency, interference, appraisal of distress), self-efficacy, and barriers to self-management. Patient Outcomes: Quality of life, anxiety and depression will be assessed at baseline and weeks 4, 8, and 12. The investigators predict that the COPE group will show significant improvement in depression, anxiety, quality of life, symptom intensity, distress, frequency and interference, self-efficacy, and perceived barriers to care, as well as decreased utilization of health care resources compared with the two control groups. Data will be analyzed using repeated measures multivariate analysis of variance using a mixed model approach.

ELIGIBILITY:
Inclusion Criteria:

* Breast, colorectal, lung or prostate cancer patients with baseline scores on intensity, distress, and/or interference => 4 on at least 2 symptoms
* Literate in English
* Must pass mental status screening and functional status at the level of ECOG 3 or lower

Exclusion Criteria:

* patients who plan to leave Florida during the summer,
* are in hospice care, or
* confused, or
* expected to die within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Quality of Life (The Multidimensional Quality of Life scale) | 13 weeks
  The Multidimensional Quality of Life scale - Cancer will be used to assess the patient's health-related quality of life
Anxiety (State-Trait Anxiety Inventory) | 13 weeks
  State Anxiety will be assessed using the State-Trait Anxiety Inventory.
Depression (The Centers for Epidemiologic Study - Depression) | 13 weeks
  The Centers for Epidemiologic Study - Depression will be used to measure depressive symptoms.

SECONDARY OUTCOMES:
Health Services Utilization (The Health Services Utilization Index) | 13 weeks
  The Health Services Utilization Index will be used to evaluate the extent to which patients seek care at the Cancer Center versus community emergency rooms.

CONTACTS AND LOCATIONS:
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States